CLINICAL TRIAL: NCT02784431
Title: Pilot Study of the Contour Neurovascular SystemTM
Status: Terminated | Type: Interventional
Why Stopped: To obtain clinical data in EU for CE Mark
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNX065.A
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Intracranial Aneurysm
Keywords: Brain; Intracranial Aneurysm Treatment; Endovascular Treatment; Brain Aneurysm; Neurovascular diseases; Aneurysms; Cerebrovascular Disorders; Central Nervous System Diseases; Vascular diseases
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Cerebrovascular Disorders; Central Nervous System Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- Contour Neurovascular System placement (Experimental): Treatment of intracranial aneurysm with the Contour Neurovascular System device.
  Interventions: Device: Contour Neurovascular System placement

INTERVENTIONS:
Device: Contour Neurovascular System placement — Patients who meet the eligibility criteria will have their target aneurysm treated with the Contour Neurovascular System device via standard endovascular procedure.

SUMMARY:
Prospective, single arm, multi centre study to evaluate the safety and performance of the Contour Neurovascular SystemTM in the treatment of intracranial aneurysm (IA)

DETAILED DESCRIPTION:
Prospective, single-arm, multi-centre European study to evaluate the safety and performance of the Contour Neurovascular SystemTM in the treatment of intracranial aneurysm (IA). Target aneurysms are unruptured aneurysms requiring endovascular treatment in the anterior and posterior cerebral circulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years at screening
2. Unruptured saccular IA in the anterior or posterior circulation with dimensions consistent with Table 2
3. IA appears suitable for Contour Neurovascular SystemTM device Patient has the necessary mental capacity to participate and is willing and able to participate in the study for the duration of the study follow-up and is able to comply with study requirements Patient able to understand and sign a study-specific informed consent form

Exclusion Criteria:

1. Ruptured IA
2. Any other IA that requires treatment in the next year
3. IA width >8.5 or <2 mm
4. IA neck >8 or <2 mm
5. IA minimum height <4mm
6. IA embolisation would most likely cause stroke
7. Target IA contains other devices/implants (e.g., coils)
8. Inability to access the target IA with the microcatheter
9. Any congenital or iatrogenic coagulopathy
10. Platelet count <50,000/microliter
11. Known allergy to platinum, nickel or titanium
12. Known allergy to contrast agents
13. Stenosis of the target IA's parent vessel >50%
14. Taking daily aspirin or other platelet inhibitor (clopidogrel or equivalent) other than for the target aneurysm
15. Taking any anticoagulants (e.g., warfarin)
16. Abnormal clotting parameters
17. Pregnant, breastfeeding or planning pregnancy in the next 2 years
18. Other medical conditions that could increase the risk of neurovascular procedures (e.g., liver failure, cancer, etc.) or ability to comply with study requirements Participating in another study with investigational devices or drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated: Patients who met the eligibility criteria and underwent an treatment attempt with the Contour Neurovascular System.
Period: Overall Study
Arm/Group | Treated
Started | 20
Completed | 0
Not Completed | 20
Not completed — Unsuccessful Implant Attempt | 1
Not completed — Early Study Termination | 19

BASELINE CHARACTERISTICS:
Arm/Group | Treated
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [43.4 to 74.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Asian | 2
  Turkish | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 18
  Hungary | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Major Ipsilateral Stroke/SAH or Death Due to Neurologic Cause Within Six (6) Months After Treatment.
Description: Percentage of subjects with major ipsilateral stroke/SAH or death due to neurologic cause within six (6) months after treatment. All neurological events were adjudicated by an independent Medical Monitor.
Time Frame: 6 months
Population: Patients who were successfully implanted with the Contour device.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 19
Participants | 0

2. Secondary Outcome: Occlusion Status of the Target IA
Description: Last known occlusion status of the target IA as judged by an independent core laboratory using the Raymond-Roy occlusion scale (Class 1 - Complete occlusion; Class 2 - Residual neck; Class 3 - Residual aneurysm).
Time Frame: 6 months (3 patients), 1 year (14 patients), 2 year (2 patients)
Population: Patients successfully implanted with the Contour device.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 19
Participants
  Class 1 | 11
  Class 2 | 3
  Class 3 | 5

ADVERSE EVENTS:
Time Frame: 1 year (9 patients), 6 months (5 patients), 6 weeks (4 patients), hospital discharge following index procedure (1 patient).
Arm/Group | Treated
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated (N=19)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Other - Unrelated to device or procedure (General disorders) | 2 (2)
Device deployment issue (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated (N=19)
Headache (Nervous system disorders) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Other - Not related to device or procedure (General disorders) | 9 (19)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor due to slow enrollment and a change in regulatory strategy. Less than 50% of the planned sample size was enrolled and none of the subjects had been followed for the planned 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02784431/Prot_SAP_000.pdf